CLINICAL TRIAL: NCT00181246
Title: Efficacy of Transdermal Fentanyl for Chronic Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20021288
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Peripheral Neuropathy; Complex Regional Pain Syndromes (CRPS)
Keywords: Neuropathic pain; Efficacy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Complex Regional Pain Syndromes; Neuralgia

INTERVENTIONS:
Drug: Transdermal Fentanyl

SUMMARY:
The efficacy of fentanyl TTS for the treatment of neuropathic pain remains to be established, although opioids in general are clearly effective for neuropathic pain and fentanyl TTS has been shown to be effective for treating other types of pain. We propose to measure functional outcomes, pain relief and side effects of fentanyl TTS for the treatment of neuropathic pain. Measures will be made at baseline and after titrating the drug to an effective level.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Neuropathic pain persisting for > 3 months
* Pain over the immediate previous three months
* The average of the least and usual pain intensity rating of 3 or greater (0-10 numerical rating scale) during the last week prior to enrollment

Exclusion Criteria:

* A history of substance abuse
* Allergic reaction to an opioid
* Significant pain of alternate etiology other than the neuropathic pain state
* Severe pulmonary disease
* Recent myocardial infarction (within the preceding three months)
* Pregnancy
* Dementia
* Encephalopathy
* Those with life expectancy of less than six months and HIV seropositivity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53
Dates: Start 2003-10; Study Completion 2005-09

PRIMARY OUTCOMES:
Change in pain intensity (0-10) and daily activity

SECONDARY OUTCOMES:
Pain relief (0-100%)
Cognition (digital symbol and grooved peg-board)
Impairment of function (MPI) and affect (BDI)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasa N Raja, MD, Principal Investigator — Johns Hopkins University